| _ | |
|---------------|----|
| $\overline{}$ | |
| ш | |
| | ۰ |
| | • |
| $\subset$ | ۰ |
| $\subset$ | |
| $\subset$ | |
| 0 | |
| $\sim$ | |
| ( | |
| $\subset$ | |
| 0 | ı |
| | • |
| ū | |
| П | |
| ~ | |
| - 1 | |
| Δ | |
| C | |
| 11 | |
| - | |
| ( | |
| - 1 | |
| d | ٠ |
| Ц | ۰ |
| | ۰ |
| _ | • |
| . 1 | |
| $\Gamma$ | |
| ~ | |
| • | |
| _ | |
| - 1 | |
| | į, |
| 0 | • |
| = | |
| ( | • |
| - | • |
| ш | |
| _ | |

| Sponsor: | BIOTRONIK SE & Co. KG |
|---|---|
| Study name / EAC code: | BIO Sync-HUTT / BA117 |
| Version and date of the<br>Statistical Analysis Plan: | 1-0, dated 15-Sept-2023 |
| Version and date of the underlying Clinical Investigation Plan: | 2-0, dated 20-Apr-2022 |

| Print Name & Title | Signature | Date of Signature<br>(DD MMM YYYY) |
|--------------------|-----------|------------------------------------|
| | | 15 SEP 2023 |
| | | 15-SEP-2023 |

# **Table of Content**

| Table of Content 1 Change History | 2 | |
|---|---|---|
| Version 1.0 | | 2 |
| | 4 | J |
| | · | 1 |
| 2.1 Aim | 4 | 4 |
| 2.2 Data for which quality control is required | 4 | 4 |
| 2.3 Unblinding | 4 | 4 |
| 2.4 General information | | 5 |
| 3 Clinical Investigation | 6 | _ |
| 3.1 Objective(s) | ( | 6 |
| 3.2 Investigational device | | 6 |
| 3.3 Design & time course | ( | 6 |
| 4 Data source | 8 | |
| 5 General statistical procedures | 8 | |
| 6 Analysis set(s) and other global variables | 10 | |
| 6.1 Analysis set of enrolled patients | 10 | 0 |
| 7 Analyses: Baseline | 10 | |
| 7.1 Analysis set | 10 | 0 |
| 7.2 Variables | 10 | 0 |
| Baseline / Demographics | 10 | C |
| Baseline / Previous Tilt test | 10 | |
| Baseline / ECG diagnostics | 1: | |
| Baseline / Syncope and pre-syncope questionnaires | 12 | |
| Medical history / Known Cardiac History - Heart Diseases | 13 | |
| Medical history / Known Cardiac History - Brady- and Tachyarrhythmias | 14 | |
| 7.3 Missing, unused or spurious data | 20 | |
| 7.4 Hypotheses & statistical tests | 20 | |
| 8 Analyses: Data of interest | 20 | _ |
| 9 Abbreviations | 24 | |
| | ۷+ | |

# **1 Change History**

Version 1.0

Initial document.



# 2 Introduction

# 2.1 Aim

The aim of this document is to provide detailed instructions on statistical analyses for the Clinical Investigation Report (CIR).

# 2.2 Data for which quality control is required

A quality control is needed for analyses of all data of interest as defined in the clinical investigation plan (CIP).

# 2.3 Unblinding

Not applicable.



# 2.4 General information

This SAP may contain verbatim excerpts from the version of the CIP specified at the cover sheet. Such excerpts are *italicized with light blue background*.

The main aspects and the design of the clinical investigation are presented in chapters 3-4.

General statistical procedures are summarized in chapter 5. Those methods are used in case there is no other specification within this document.

Analysis set(s) and other global variables are defined in detail in chapter 6.

Descriptive and inferential statistical analyses for endpoint(s) are handled in following chapters. Thereby the following statistical considerations are specified:

- Analysis set: Definition of the analysis population (e.g. Intention-to-Treat or Per-Protocol for controlled clinical investigations or all patients with valid informed consent for singlearm clinical investigations)
- Variable characteristics: Description of all relevant variables (directly addressable from validated tools, e.g. CDMS or CDW, and derived variables) such as variable name, variable label, variable values, and data type.
- Derived variables, if applicable: For variables, which are not directly addressable from validated tools but are derived from other variables, pseudo-code or other instructions for the variable construction shall be provided.
- Missing, unused or spurious data: Specification of all data to be excluded from the specific analysis, e.g. data measured after a pre-specified point in time or implantation date after pre-hospital discharge date; specification whether and -if applicable- how to impute missing data.
- Data analysis: Description of descriptive, exploratory, and confirmatory analyses in text, tables, or pseudo-code shall be provided for unambiguous data analysis.

All variables are defined in tables using the following columns:

Data file: Name of a data file exported from the CDMS and unique identifier, if applicable (e.g. patient-specific "patient\_display\_ID\_full" or event-specific record\_ID); new data files ("data\_SAR") may be generated by merging all relevant data from the original CDMS data files and generating derived variables;

Notes: Information whether data shall be presented with "descriptive" methods as defined in this SAP, data for "case listings" of original data for each patient specified, or "no report" for data needed for generating derived variables only;

Variable name: Original name of CDMS data or new name of a derived variables (indicated with a prefix "SAR\_" or a suffix "\_SAR");

Variable label: Original labels of CDMS data will be used for generating the SAR unless a new label is defined in this document ("NEW");

Variable level: Nominal, ordinal, scale (synonymous for metric, continuous, interval scale and/or ratio scale), or date;

Nominal values: Original values of CDMS of nominal or ordinal data will be used unless new values are defined in this document ("NEW").

| Data file, | Notes | Variable | Variable | Variable | Nominal values |
|---|---|---|---|---|---|
| identifier | | name | label | level | |
| patient_display_id_full | | | | | |



# 3 Clinical Investigation

# 3.1 Objective(s)

# CIP chapter 7.1

The purpose of this study is to add knowledge to better understand the hemodynamic mechanisms underlying recurrent syncopal events and optimal pacing programming.

## CIP chapter 7.2

This study will provide standardized, complete and quality controlled data sets with parameters that describe hemodynamic changes and their timing with respect to CLS pacing activation during reflex syncope induced by HUTT.

# 3.2 Investigational device

# CIP chapter 4 Device(s) used in the study

The following devices, tools and accessories will be used during the study:

 the CLS algorithm (as investigational device in this investigation according to, ISO14155) implemented in current dual-chamber pacemakers manufactured by:

BIOTRONIK SE & Co. KG

Woermannkehre 1

12359 Berlin

Germany

www.biotronik.com

- RENAMIC programmers or later models;
- Any external monitor capable of measuring continuously patient's hemodynamics (e.g. Task Force Monitor);
- Standard equipment needed for the HUTT execution.

Such devices must be available at the investigational sites before study participation and will not be provided by the Sponsor.

# 3.3 Design & time course

# CIP chapter 8.1.1

The study is designed as a prospective, non-randomized, multi-center, observational acute study without additional follow-ups after HUTT execution.

# CIP chapter 8.2.4 Point of enrollment

A subject is considered enrolled in the BIO\Sync-HUTT Study upon the signature of the Informed Consent Form after confirmation of the elegibility criteria by the investigator.

# CIP chapter 8.2.6 Expected duration of each subject's participation

Subjects participate from consent to HUTT execution with not further follow-up.

CIP chapter 9.1 Overview (study procedures)



This section describes all the study-related procedures as listed in Table 1 which will be performed during a routine scheduled patient follow-up. Prior to obtaining informed consent, the patient's background and medical history will be reviewed in order to ensure he/she is an appropriate candidate for the study. Patient who undergo HUTT during ordinary follow-up visits irrespective of study participation, is eligible. After the patient has been determined to be eligible for the study, written informed consent will be obtained and demographic and medication data will be collected. Syncope and presyncope questionnaires will be self-administered. Prior to the HUTT, pacemaker interrogation will be performed in order to check programming settings and to collect device diagnostics. The HUTT may be performed and also recorded by a high-definition camera if available. Full hemodynamic parameters and ECG traces will be acquired during the HUTT. Any collected data and adverse events will be documented in an electronic CRF.

| Investigations | Enrollment/study visit |
|---|---|
| Verification of in- and exclusion criteria | Х |
| Patient informed consent | X |
| Demographic data | X |
| Medical history | Χ |
| Co-morbidities | X |
| Medication therapy | X |
| Patient self-administered syncope and pre-syncope questionnaires | Х |
| ECG | X |
| Device programming settings and diagnostics | X |
| Head-up tilt test (including video recording if available) | Х |
| Collection of primary and secondary endpoint-related measurements | Х |
| (S)AE, (S)ADE, DD monitoring | Χ |

# 4 Data source

All the following datasets are exported from the CDMS:

- Enrollment
- Baseline
- Medical History
- Device Log
- Device Interrogation
- HUTT
- Study Termination
- Adverse Event
- Device Deficiency
- Deviation (patient related)

All datasets except "adverse\_event" and "device\_log\_details" are patient-specific, i.e. one data row per patient.

# 5 General statistical procedures

CIP chapter 12 Statistical Design and Analysis

12.2 Descriptive statistics

Standard descriptive statistical methods are used depending on the type of the available data. For continuous variables, mean value, standard deviation, median, minimum, maximum and quartiles are calculated. For nominal variables, absolute and relative frequencies are calculated based on non-missing data. For ordinal variables, median, minimum, maximum and quartiles or absolute and relative frequencies are calculated for each category based on non-missing data. Shapiro-wilk test for normality for each variable is used.

# 12.3 Analytical procedures

Standard inferential statistical methods may be used depending on the type of the available data. For mean values, confidence intervals are calculated based on a t-distribution. For relative frequencies, confidence intervals are calculated based on a binomial distribution. Thereby, the significance value specified in the following sub-chapter is considered.

# 12.4 Significance level, statistical power, and statistical testing

This document and/or its contents are only for internal use.

Because there are no pre-specified hypotheses, all analyses are exploratory. However, a result of a two-sided statistical test with a p-value less than 5% or a one-sided statistical test with a p-value less than 2.5% is considered statistically significant.

For any inferential analyses, the result of a two-sided statistical test with a p-value less than 5% or a one-sided statistical test with a p-value less than 2.5% is considered statistically significant.

# 12.6 Interim analyses





There are no pre-planned interim analyses.

### 12.7 Bias

In case of a clear evidence of bias, which was not considered before, the Statistical Analysis Plan (SAP) is updated to avoid any bias.

# 12.10 Confounding factors (CIP chapter 8.1.2 Measures taken to minimize or avoid bias)

Accurate patient selection as described in section 8.2 and precise conduction of HUTT according to the procedures described in section 9 will allow to minimize potential confounding factors.

# 12.9 Missing, unused, and spurious data

All data needed to be analyzed are pre-documented in a Statistical Analysis Plan (SAP).

During a blind review process before any pre-planned analysis, missing and spurious data, which are relevant at least for the endpoints, are identified. In case such data can't be clarified via a query management process, the Statistical Analysis Plan (SAP) is updated to avoid any bias. If appropriate, analyses will be performed both with/without spurious data. Number of missing data are reported for each descriptive and inferential analysis in the Statistical Analysis Report (SAR) and Clinical Investigation Report (CIR), if applicable. Spurious data are commented in the Clinical Investigation Report (CIR), if applicable. Drop-outs are reported in the Statistical Analysis Report (SAR) and Clinical Investigation Report (CIR), if applicable. Missing data will not be replaced.

# 12.14 Exploratory analysis and sensitivity analysis Not applicable.

# 12.15 Deviations from the original statistical plan

A Statistical Analysis Plan (SAP) is provided after go-life of the Clinical Data Management System (CDMS). The SAP can be updated before CDMS-freeze or closure based on a review of the data, whereby the new version is containing a change history. Any deviation from the valid SAP version with respect to inferential analyses are indicated in the Clinical Investigation Report (CIR), if applicable.

# 6 Analysis set(s) and other global variables

# 6.1 Analysis set of enrolled patients

CIP chapter 12 Statistical Design and Analysis

13.1 Analysis population

All patients with valid patient informed consent (ICF) are included in the analysis set.

# 7 Analyses: Baseline

# 7.1 Analysis set

All analyses are performed for the analysis set with valid informed consent.

# 7.2 Variables

# Baseline / Demographics

| Data file, | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| baseline | descriptive | dmsex | Gender | nominal | ∘ Yes ∘ No |
| | descriptive | dmage | Age [Years] | scale | n.a. |



# Baseline / Previous Tilt test

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| Baseline | descriptive | QSHUR | Response to tilt test | nominal | ∘ Syncope<br>∘ Pre-syncope |
| Baseline | descriptive | QSHURF | Response phase of the tilt test | nominal | <ul> <li>Positive during passive<br/>phase</li> <li>Positive after nitroglycerin<br/>(TNT) administration</li> </ul> |
| baseline | descriptive | EGHUTYP | Type of electrocardiographic manifestation induced by tilt testing | nominal | <ul><li>Sinus arrest</li><li>Atrioventricular block</li><li>Other</li></ul> |



| baseline | Case listing | COHUTYP | Specification of other | text | o <b>n.a.</b> |
|---|---|---|---|---|---|
| | for | | type of | | |
| | EGHUTYP = | | electrocardiographic | | |
| | Other | | manifestation induced | | |
| | | | by tilt testing | | |
| Baseline | Descriptive | EGMASPU | Maximum asystolic | scale | o <b>n.a.</b> |
| | | | pause [s] | | |



# Baseline / ECG diagnostics

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| baseline | descriptive | | Atrial rhythm during ECG recording | nominal | <ul> <li>Sinus rhythm</li> <li>Atrial fibrillation</li> <li>Atrial flutter/other SVT</li> <li>Atrial paced rhythm</li> <li>Other</li> </ul> |
| baseline | Case listing<br>for<br>CVEGARH =<br>Other | COEGARH | Specification of other atrial rhythm during ECG recording | Text | n.a. |
| baseline | descriptive | CVEGVRH | Ventricular rhythm<br>during ECG recording | nominal | o Intrinsic - atrial<br>conducted<br>o Intrinsic - escape rhythm<br>o Ventricular paced rhythm<br>o Other |



| baseline | Case listing<br>for CVEGVRH<br>= Other | COEGVRH | Specification of other ventricular rhythm during ECG recording | Text | n.a. |
|---|---|---|---|---|---|
| baseline | descriptive | EGHRTR | Resting HR [bpm] | scale | n.a. |
| baseline | descriptive | EGPRI | PR interval [ms] | scale | n.a. |
| baseline | descriptive | QSEGABN | Any relevant findings in resting ECG? | nominal | ∘ Yes ∘ No |
| baseline | Case listing<br>for QSEGABN<br>= Yes | COEGABN | Specification of relevant findings | Text | n.a. |

# Baseline / Echocardiography diagnostics

| Data file,<br>identifier<br>patient_<br>display_id_full | | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|
| baseline | descriptive | Left ventricular ejection [%] | Scale | n.a. |



# Baseline / Syncope and pre-syncope questionnaires



| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| baseline | descriptive | CESNC | Have you experienced episodes of syncope and/or pre-syncope after the pacemaker implantation? | nominal | ∘ Yes ∘ No |
| baseline | Descriptive<br>for CESNC =<br>Yes | CESNCTOT | Total number of syncope/s | Scale | n.a. |
| baseline | Descriptive<br>for CESNC =<br>Yes | CEPSNCTO | Total number of pre-syncope/s | Scale | n.a. |



# Medical history / Known Cardiac History - Heart Diseases

| Data file, identifier patient_display_id_full | Notes | Variable<br>name | Variable<br>label | | Nominal<br>values |
|---|---|---|---|---|---|
| medical_ | descriptive | MHHF | History of heart failure | nominal | ∘ Yes ∘ No |
| history | | MHCAD | History of coronary artery disease | nominal | ∘ Yes ∘ No |
| | | MHHHD | Hypertensive heart disease | nominal | ∘ Yes ∘ No |
| | | MHVHD | Valvular heart disease | nominal | ∘ Yes ∘ No |
| | | MHHCM | Hypertrophic cardiomyopathy | nominal | ∘ Yes ∘ No |
| | | MHRCM | Restrictive cardiomyopathy | nominal | ∘ Yes ∘ No |
| | | MHDCM | Dilated cardiomyopathy | nominal | ∘ Yes ∘ No |
| | | MHHDOTH | Other heart diseases | nominal | ∘ Yes ∘ No |
| medical_<br>history | Case listing for MHHDOTH = Yes | COHDOTH | Specification of other heart diseases | Text | n.a. |



All rights pertaining to this document are exclusively held by BIOTRONIK SE & Co. KG. Any non-authorized copying, reproduction or distribution is not permitted. Confidentiality: This document and/or its contents are only for internal use.





# Medical history / Known Cardiac History - Brady- and Tachyarrhythmias

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| medical_<br>history | descriptive | MHAVB | History of AV block | Nominal | o Yes<br>o No |
| medical_<br>history | Descriptive<br>for<br>MHBBBTYP =<br>Yes | MHAVBTYP | Type of AV block | Nominal | o AV block I°<br>o AV block II°<br>o AV block III° |
| medical_<br>history | descriptive | МНВВВ | History of bundle<br>branch block | nominal | o Yes<br>o No |
| medical_<br>history | Descriptive<br>for MHBBB =<br>Yes | MHBBBTYP | Type of bundle<br>branch block | nominal | o LBBB<br>o RBBB<br>o Other |
| medical_<br>history | Case listing<br>for<br>MHBBBTYP =<br>Other | COBBBTYP | Specification of other type of bundle branch block | Text | n.a. |
| medical_<br>history | descriptive | MHCNDDOT | History of other type of conduction disease | nominal | o Yes<br>o No |





| medical_<br>history | Case listing for MHCNDDOT = Yes | COCNDDOT | Specification of other type of conduction disease | Text | n.a. |
|---|---|---|---|---|---|
| medical_<br>history | descriptive | MHAFB | History of atrial fibrillation | nominal | o Yes<br>o No |
| medical_<br>history | Descriptive<br>for MHAFB =<br>Yes | CVAFBTYP | Type of atrial fibrillation | nominal | o Paroxysmal<br>o Persistent<br>o Long-standing persistent<br>o Permanent |
| medical_<br>history | descriptive | MHAVA | History of other atrial/supraventricular arrhythmias | nominal | o Yes<br>o No |
| medical_<br>history | Descriptive<br>for MHAVA =<br>Yes | MHAFL | History of atrial flutter | nominal | o Yes<br>o No |
| medical_<br>history | Descriptive<br>for MHAVA =<br>Yes | MHAT | History of atrial tachycardia | nominal | o Yes<br>o No |
| medical_<br>history | Descriptive<br>for MHAVA =<br>Yes | MHSVT | History of supraventricular tachycardia | nominal | o Yes<br>o No |
| medical_<br>history | Descriptive<br>for MHAVA =<br>Yes | MHAVAOTH | History of other type of atrial/ supraventricular arrhythmias | nominal | o Yes<br>o No |
| medical_<br>history | Case listing for MHAVAOTH = Yes | COAVAOTH | Specification of other type of atrial/ supraventricular arrhythmias | Text | n.a. |
| medical_<br>history | descriptive | MHVA | History of ventricular arrhythmias | nominal | o Yes<br>o No |
| medical_<br>history | Case listing<br>for MHVA =<br>Yes | COVA | Specification of ventricular arrhythmias | Text | n.a. |











# Medical history / Known Co-morbidities

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| medical_<br>history | descriptive | MHHP | Hypertension (including well-controlled) | nominal | o Yes<br>o No |
| medical_<br>history | descriptive | MHASTH | Asthma or other chronic lung disease (except COPD) | nominal | o Yes<br>o No |
| medical_<br>history | descriptive | MHCOPD | Chronic obstructive pulmonary disease (COPD) | nominal | o Yes<br>o No |
| medical_<br>history | descriptive | MHCKD | Chronic renal<br>insufficiency / chronic<br>kidney disease (CKD)<br>(i.e. eGFR < 60<br>ml/min/1.73 m <sup>2</sup> ) | nominal | o Yes<br>o No |
| medical_<br>history | descriptive | MHDIAM | Diabetes mellitus | nominal | o Yes<br>o No |
| medical_<br>history | descriptive | MHNEUD | Neurological disease | nominal | o Yes<br>o No |
| medical_<br>history | descriptive | MHCNCR | Cancer | nominal | o Yes<br>o No |
| medical_<br>history | descriptive | MHHPLP | Hyperlipidemia | nominal | o Yes<br>o No |
| medical_<br>history | descriptive | МНСМВОТН | Other co-morbidities | nominal | o Yes<br>o No |
| medical_<br>history | Case listing<br>for<br>MHCMBOTH<br>= Yes | СОСМВОТН | Specification of other co-morbidities | Text | n.a. |









# Medical history / Medication therapy

| Data file,<br>identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | Variable<br>label | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| medical_<br>history | descriptive | CMCVM01 | ACE inhibitors | nominal | o Yes<br>o No |
| | descriptive | CMCVM02 | Angiotensin II receptor blocker | nominal | o Yes<br>o No |
| | descriptive | CMCVM03 | Ca2 antagonist | nominal | o Yes<br>o No |
| | descriptive | CMCVM04 | Alpha – Antagonist | nominal | o Yes<br>o No |
| | descriptive | CMCVM05 | Beta blocker | nominal | o Yes<br>o No |
| | descriptive | CMCVM06 | Diuretics including aldosterone blocker | nominal | o Yes<br>o No |
| | descriptive | CMCVM07 | Antiarrhythmic drugs | nominal | o Yes<br>o No |
| | Descriptive<br>for CMCVM07<br>= Yes | CMCVM08 | Sotalol | nominal | o Yes<br>o No |



| , CRQ200005199 |
|------------------------------------|
| FOR-137- 059-C / SOP-137-060.020 / |

| for CMCVM07 | CMCVM09 | Amiodarone | nominal | o Yes<br>o No |
|---|---|---|---|---|
| = Yes Descriptive for CMCVM07 = Yes | CMCVM10 | Other antiarrhythmics | nominal | o Yes<br>o No |
| | COCVM10 | Specification of Other antiarrhythmics | Text | n.a. |
| descriptive | CMCVM11 | Anticoagulants | nominal | o Yes<br>o No |
| Case listing for CMCVM11 = Yes | COCVM11 | Specification of anticoagulants | Text | n.a. |
| descriptive | CMCVM12 | Antiplatelet agents | nominal | o Yes<br>o No |
| descriptive | CMCVM13 | NSAIDs (nonsteroidal anti-inflammatory drugs) | nominal | o Yes<br>o No |
| descriptive | CMCVM14 | Vasodilator agents | nominal | o Yes<br>o No |
| descriptive | CMCVM15 | Nitrates | nominal | o Yes<br>o No |
| descriptive | CMCVM16 | Digitalis | nominal | o Yes<br>o No |
| descriptive | CMCVM17 | Lipid lowering agents | nominal | o Yes<br>o No |
| Case listing for CMCVM17 = Yes | COCVM17 | Specification of lipid lowering agents | Text | n.a. |
| descriptive | CMCVM18 | Psychiatric drugs | nominal | o Yes<br>o No |
| descriptive | CMCVMOTH | Other | nominal | o Yes<br>o No |
| Case listing for CMCVMOTH = Yes | COCVMOTH | Specification of other | text | n.a. |











# 7.3 Missing, unused or spurious data

See chapter 5.

# 7.4 Hypotheses & statistical tests

There are no pre-defined statistical hypotheses.

# 8 Analyses: Data of interest

All analyses are performed for the enrollment analysis set with valid informed consent and DDD-CLS pacing mode activated according to the CIP.

# 10.1 Study-specific dates

| Data file: | Notes | Variable | Variable | Variable | Nominal |
|---|---|---|---|---|---|
| Identifier | | name | label | level | values |
| patient_ | | | | | |
| display_id_full | | | | | |
| device_log_det | No report | PRIMSTDT | Implantation/Use date | date | n.a. |
| ails | - | | | | |
| hutt | No report | SVHUSTDT | Date of visit | date | n.a. |
| Data_SAR | Descriptive | TIME_IMPL_HUTT | Days from implantation to HUTT | Scale | n.a. |
| | | _SAR | examination [years] | | |



# 10.2 HUTT

| Data file:<br>Identifier<br>patient_<br>display_id_full | Notes | Variable<br>name | | Variable<br>level | Nominal<br>values |
|---|---|---|---|---|---|
| hutt | Case listing | CVMHRTTM | Time of maximum spontaneous heart rate (end of phase 1/beginning phase 2 of the reflex) | Scale | n.a. |
| | descriptive | QSHUPMPC | Did the pacemaker pace during HUTT? | nominal | o Yes<br>o No |
| | Case listing | PRPCSTTM | Time of pacing onset/maximum pacing rate | scale | n.a. |
| | Case listing | PRHRPCTM | Time of recovery of basic pacing rate or spontaneous rhythm after pacing (end of recovery period) | Scale | n.a. |
| | Case listing | PRHRHRTM | Time of recovery of starting spontaneous heart rate | Scale | n.a. |



| _ | ı |
|---------------|---|
| U | 3 |
| σ | ٦ |
| ÷ | 4 |
| 10 | ١ |
| 7 | ś |
| č | ζ |
| | 2 |
| $\subset$ | J |
| $\subset$ | כ |
| 0 | J |
| r | ۱ |
| | , |
| Ö | - |
| L | J |
| _ | • |
| $\overline{}$ | 2 |
| | , |
| $\overline{}$ | V |
| $\subset$ | כ |
| c | : |
| 4 | 2 |
| Ū | כ |
| $\subset$ | ٥ |
| - 1 | |
| $\vdash$ | • |
| ~ | ٦ |
| - | Á |
| 'n | |
| ۵ | |
| | 5 |
| C | , |
| U | ) |
| - | ` |
| ( | ) |
| ٦ | • |
| ά | ١ |
| ŭ | |
| 느 | 2 |
| _ | ) |
| ĸ. | L |
| `~ | j |
| ٠. | |
| _ | 1 |
| J | , |
| Ω | _ |
| $\overline{}$ | ١ |
| ĭ | • |

| | (for QSHUPMPC<br>= No) | | | |
|---|---|---|---|---|
| descriptive | QSHÚSNC | Did syncope (i.e. loss of consciousness) occur during HUTT? | Nominal | n.a. |
| Case listing | QSSNCTM | Time of syncope | Scale | n.a. |
| Case listing | QSTDTM | Time of tilt-down (supine patient position just after tilt-down) | scale | n.a. |
| descriptive | QSHRHRDU | Duration of the recovery phase (interval from maximum pacing rate to basic rate or spontaneous rhythm from the start of the HUTT) [sec] | Scale | n.a. |
| descriptive | CVHRHUST | HR at HUTT start [bpm] (upright patient position just after tilt) | Scale | n.a. |
| descriptive | CVMHRT | HR at time of maximum spontaneous heart rate (end of phase 1/beginning phase 2 of the reflex) [bpm] | Scale | n.a. |
| descriptive | CVHRPC | HR at time of pacing onset/maximum pacing rate [bpm] | Scale | n.a. |
| descriptive | CVHRAPC | HR at time of recovery of basic pacing rate or spontaneous rhythm after pacing (end of recovery period) [bpm] | Scale | n.a. |
| descriptive | CVHRAPCN | HR at time of recovery of basic pacing rate or spontaneous rhythm after pacing not applicable | | o True<br>o False |
| descriptive | CVHRHU | HR at time of syncope during HUTT [bpm] | Scale | n.a. |
| descriptive | CVHRAHU | HR at time of tilt-down | Scale | n.a. |
| descriptive | CVSBPHST | Systolic BP at HUTT start [mmHg] | Scale | n.a. |
| descriptive | CVDBPHST | Diastolic BP at HUTT start [mmHg] | Scale | n.a. |
| descriptive | CVSBPMHR | Systolic BP at time of maximum spontaneous heart rate (end of phase 1/beginning phase 2 of the reflex) [mmHg] | Scale | n.a. |
| descriptive | CVDBPMHR | Diastolic BP at time of maximum spontaneous heart rate (end of phase 1/beginning phase 2 of the reflex) [mmHg] | Scale | n.a. |
| descriptive | CVSBPPC | Systolic BP at time of pacing onset/maximum pacing rate [mmHg] | Scale | n.a. |
| descriptive | CVDBPPC | Diastolic BP at time of pacing onset/maximum pacing rate [mmHg] | Scale | n.a. |
| descriptive | CVSBPAPC | Systolic BP at time of recovery of basic pacing rate or spontaneous rhythm after pacing (end of recovery period) [mmHg] | Scale | n.a. |
| descriptive | CVDBPAPC | Diastolic BP at time of recovery of basic pacing rate or spontaneous rhythm after pacing (end of recovery period) [mmHg] | Scale | n.a. |
| descriptive | CVSBPHU | | Scale | n.a. |
| descriptive | CVDBPHU | Diastolic BP at time of syncope during HUTT [mmHg] | Scale | n.a. |
| descriptive | CVSBPAHU | Systolic BP at time of tilt-down (supine patient position just after tilt-down) [mmHg] | Scale | n.a. |
| descriptive | CVDBPAHU | Diastolic BP at time of tilt-down (supine patient position just after tilt-down) [mmHg] | Scale | n.a. |



| , CRQ200005199 |
|------------------------------------|
| FOR-137- 059-C / SOP-137-060.020 / |

| | descriptive | CVSVHUST | SV at HUTT start [ml] | Scale | n.a. |
|---|---|---|---|---|---|
| | descriptive | CVSVMHRT | SV at time of maximum spontaneous heart rate (end of phase 1/beginning phase 2 of the reflex) [ml] | Scale | n.a. |
| descriptive | | CVSVPC | SV at time of pacing onset/maximum pacing rate [ml] | Scale | n.a. |
| | descriptive | CVSVAPC | SV at time of recovery of basic pacing rate or spontaneous rhythm after pacing (end of recovery period) [ml] | Scale | n.a. |
| | descriptive | CVSVHU | SV at time of syncope during HUTT [ml] | Scale | n.a. |
| | descriptive | CVSVAHU | SV at time of tilt-down (supine patient position just after tilt-down) [ml] | Scale | n.a. |
| | descriptive | CVTPRHUS | TPR at HUTT start [dyn·s/cm5] | Scale | n.a. |
| | descriptive | CVTPRMHR | TPR at time of maximum spontaneous heart rate (end of phase 1/beginning phase 2 of the reflex) [dyn·s/cm5] | Scale | n.a. |
| | descriptive | CVTPRPC | TPR at time of pacing onset/maximum pacing rate [dyn·s/cm5] | Scale | n.a. |
| | descriptive | CVTPRAPC | TPR at time of recovery of basic pacing rate or spontaneous rhythm after pacing (end of recovery period) [dyn·s/cm5] | Scale | n.a. |
| | descriptive | CVTPRHU | TPR at time of syncope during HUTT [dyn·s/cm5] | Scale | n.a. |
| | descriptive | CVTPRAHU | TPR at time of tilt-down (supine patient position just after tilt-down) [dyn·s/cm5] | Scale | n.a. |
| ermination | Case listing | COSUM | General Comments | Text | n.a. |
| ata_SAR | descriptive | SLOPE_HR_HUTT<br>_SAR | Slope in heart rate (bpm per sec) during the recovery phase | Scale | n.a. |
| ata_SAR | descriptive | SLOPE_SBP_HUT<br>T_SAR | Slope in systolic blood pressure<br>(mmHg per sec) during the<br>recovery phase | Scale | n.a. |











# 9 Abbreviations

| • | BP | Blood | pressure |
|---|----|-------|----------|
|---|----|-------|----------|

- CDMS Clinical Data Management System
- CI Confidence Interval
- CIP Clinical Investigation Plan
- CIR Clinical Investigation Report
- CLS Closed loop stimulation
- COPD Chronic obstructive pulmonary disease
- CRF Case Report Form
- CKD Chronic kidney disease
- ECG Electrocardiogram
- FU(P) Follow-up
- HR Heart Rate
- HUTT Head-up tilt test
- ICF Informed consent form
- SAP Statistical Analysis Plan
- SAR Statistical Analysis Report
- SOP Standard Operating Procedure
- SV Stroke volume
- TPR Total peripheral resistance